CLINICAL TRIAL: NCT06013891
Title: The Incidence and Association of PACU Course and Early Postoperative Complications and Deterioration
Brief Title: Observational Study of Early Postoperative Deterioration and Complications
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Lea Baunegaard Hvidberg, Clinical Nurse Specialist, Ph.d-fellow, Copenhagen University Hospital, Hvidovre
Other Study IDs: F-22045028
Record Dates: First submitted 2023-07-07; First posted 2023-08-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Complications; Deterioration, Clinical; Postoperative Care; Anesthesiology
Keywords: Postoperative Complications; Deterioration, Clinical; Postoperative Care; Clinical assessment
MeSH Terms: conditions — Postoperative Complications; Clinical Deterioration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective observational research project aims to investigate how vital sign deterioration and complications within the (PACU) relate to early deterioration and complications in the surgical wards 72 hours post-PACU discharge.

The participants studied will be high-risk surgical patients who will follow a normal postoperative course from the PACU to the surgical ward. The investigators seek to evaluate the association between deterioration and complications within the PACU with vital signs deterioration and complications in the surgical wards. Second, the investigators will explore how deterioration and complications affect PACU length of stay, morbidity, mortality, rapid response Teams call-outs (RRT) (Early warning score >7), extra medical patient supervision, and unplanned intensive care unit (ICU) admissions. The investigators will also examine the nurses' assessment of the patient's risk of deterioration and complications upon discharge from the PACU and admission to the surgical department.

DETAILED DESCRIPTION:
Postoperative complications are increasing and are an under-recognized cause of morbidity and mortality. While there has been significant attention to preoperative risk assessments for late postoperative complications and 30-day mortality, little attention has been paid to the PACU as a point of in-patient triage for early postoperative deterioration and complications. PACU to surgical ward discharge readiness is often based on a quantitative discharge score that does not account for the patient's physiological responses or distinguish between surgery type, age, and co-morbidities.

The discharge score is a clinical decision-making tool that sets the frame for the patient's readiness for discharge and functions as a "one six fits all" system. However, this "one size fits all" approach may not be adequate as a discharge tool when discharging high-risk, fragile patients from the PACU. The current evidence on using criterion-based discharge scores and the connection with early postoperative deterioration and complications are absent and need further investigation.

It is unclear whether early postoperative deterioration and complications can be predicted and assessed during PACU stay. Thus leaving a big potential for improvement in patient assessment and detection of early deterioration and complications, improving safe PACU discharge for high-risk fragile patients. Providing new knowledge on early postoperative deterioration and complications within high-risk, fragile patient groups could improve postoperative courses and patient safety.

Statistical analysis plan Data is expected to be divided into two (or 3) consecutive studies.

ELIGIBILITY:
Patients who wish to participate will sign a consent form. Baseline data will be obtained on all eligible participants; however, the full registry will only be obtained for those who permit us.

To recruit participants, the surgical schedules will be screened on a daily basis by the principal investigator and/or a member of the research team (VB).

Data entry has been prepared in RedCap, a secure method of robust data collection. All data entry will be reviewed and validated by LBH and VB. In case of discrepancies or inconsistencies, senior members of the research team NBF or EKA will review data for clarity and validation.

Inclusion Criteria:

-Adult patients undergoing surgery for a hip fracture, lower limb amputation, open liver resection, open pancreatic, and esophageal/gastric surgery

And

* Adult patients undergoing open or laparoscopic major abdominal surgery and orthopedic surgery
* Surgery time over 2 hours
* American Society of Anesthesiologists (ASA) physical status classification system 3 - 4

Exclusion Criteria:

* Pre-planned fixed minimum PACU stay
* Planned intensive care unit (ICU) stay
* Terminally ill
* Incapable of giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include approximately 250 adults undergoing surgery for hip fracture, lower limb amputation, open liver resection, open pancreatic and esophageal/gastric surgery, and open or laparoscopic major abdominal surgery. The surgical patient categories are selected based on types of surgery performed at the research sites, clinical experience, and well-known high risks of postoperative morbidity and mortality.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-03 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
The incidence of deterioration and complications during the first 72 hours post-PACU discharge and its association with deterioration and complication rates in the PACU | Up to three days
  In accordance with ICH-GCP: any untoward medical occurrence that(...)
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Requires intervention to prevent permanent impairment or damage And/or severe deviating vital signs defined as outside normal thresholds.
The incidence of deterioration and complications during PACU stay | Up to four our days
  In accordance with ICH-GCP: any untoward medical occurrence that(...)
  * Results in death
  * Is life-threatening
  * Requires inpatient hospitalization or causes prolongation of existing hospitalization
  * Results in persistent or significant disability/incapacity
  * Requires intervention to prevent permanent impairment or damage And/or severe deviating vital signs defined as outside normal thresholds.

OTHER OUTCOMES:
The association between deterioration, complications, and PACU length of stay | Up to 24 hours
  How are deterioration and/or complications associated with prolonged PACU stay PACU length of stay? (> 2 hours)
The association between individual PACU discharge score and early risk of deterioration and complications within 72 hours post-PACU discharge | Up tp 72 hours
  Can the discharge score (modified Aldrete score/aggregated score of vital signs) be a predictive value (of high individual or high total score) for early risk of deterioration and complications
The percentages of RRT call-outs (Early warning score >7) within 72 hours post-PACU discharge | Up to 72 hours post PACU discharge
  How many patients will experience an Early Warning Score >7 (Early warning score is an aggregated score of physiological parameter). At a high score of equal to or above 7, the RRT should be contacted)
The percentages of extra medical, surgical, or ICU supervision within 72 hours post-PACU discharge | Up to 72 hours post PACU discharge
  How many patients will experience extra medical, surgical, or ICU supervision within 72 hours
The percentages of unexpected patient transfer to cardiology, the pulmonary department, or the ICU | Up to four days from PACU admittance
  How many patients will experience unexpected transfer to cardiology, the pulmonary department, or the ICU
PACU nurse prediction (triage categories) of the patient course within 72 hours post-PACU discharge | At PACU discharge to surgical ward (up to 24 hours from PACU admittance)
  The triage categories are; green) stable and uncomplicated postoperative course. Yellow) Potentially unstable with a risk of minor risk of a complicated postoperative course. Orange) Unstable, at high risk of a complicated postoperative course. Red) in a critical condition with the risk off life-threatening complications
Surgical ward nurse prediction (triage categories) of the patient course within 72 hours post-PACU discharge | When the ward nurse receive the patient from the PACU (up to 24 hours of PACU admittance)
  What are the receiving ward nurse's clinical predictions of the patient course within 72 hours post-PACU discharge. The triage categories are; green) stable and uncomplicated postoperative course. Yellow) Potentially unstable with a risk of minor risk of a complicated postoperative course. Orange) Unstable, at high risk of a complicated postoperative course. Red) in a critical condition with the risk of life-threatening complications
The association between the triage categories and deterioration and complications within 72 hours post-PACU discharge | Up to 72 hours post PACU discharge or at hospital discharge (under 72 hours from PACU discharge)
  Can PACU and ward nurses predict the outcome of the patient course within the first 72 hours post PACU discharge (within the defined triage categories describing the conditions)
Agreement between the PACU nurse' and ward nurses' triage | Up to 72 hours post PACU discharge or at hospital discharge (under 72 hours from PACU discharge)
  How aligned are the PACU and ward nurses' predictions within the first 72 hours post-PACU discharge or at hospital discharge? Alignment will be explored using kappa statistics

CONTACTS AND LOCATIONS:
Overall Officials: Lea B Hvidberg, RN, Ms.c., Principal Investigator — Dep. of Anesthesiology, Amager and Hvidovre University Hospital; Eske K Aasvang, MD,Med.Sc.D., Study Chair — Centre for Cancer and Organ Diseases, Rigshospitalet, University Hospital; Martin G Tolsgaard, MD,Med.Sc.D., Study Chair — CAMES Rigshospitalet and Department of Obstetrics, Rigshospitalet, University Hospital; Nicolai B Foss, MD,Med.Sc.D., Study Chair — Department of Anesthesiology, Amager and Hvidovre University Hospital
Locations (1):
- Amager and Hviovre Universitu Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available starting 6 months after publication
Access Criteria: Data can by shared by request to the principal researcher